CLINICAL TRIAL: NCT06468969
Title: A Prospective, Single-Center, Randomized Controlled Trial Comparing Enhanced Follow-up With Standard Follow-up in Post-Gastrectomy Patients With Advanced Gastric Cancer
Brief Title: Enhanced vs. Routine Follow-Up After Total Gastrectomy for Advanced Gastric Cancer: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Support
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer; Total Gastrectomy; Postoperative Care; Quality of Life; Follow-up
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Follow-up Group (Experimental): Participants in this group will receive comprehensive follow-up care starting from the 4th week post-surgery. Every 3 weeks, they will undergo a thorough assessment that includes:
  Symptom Assessment: Comprehensive evaluation of symptoms. Nutritional Assessment: Using internationally recognized tools such as NRS 2002 and PG-SGA.
  Psychological Assessment: Utilizing tools such as the Distress Thermometer (DT), Generalized Anxiety Disorder 7-item scale (GAD-7), Fear of Cancer Recurrence 7-item scale (FCR-7), Insomnia Severity Index (ISI), and the Patient Health Questionnaire 9-item depression scale (PHQ-9).
  Interventions: Other: Enhanced Follow-up
- Standard Follow-up Group (Active Comparator): Participants in this group will receive standard postoperative follow-up care, which includes medical examinations and treatments as necessary. Nutritional and psychological assessments will only be conducted if deemed necessary by the patient or the healthcare provider. This group will serve as the control group for comparison with the enhanced follow-up group.
  Interventions: Other: Enhanced Follow-up

INTERVENTIONS:
Other: Enhanced Follow-up — Participants will receive comprehensive follow-up care starting from the 4th week post-surgery. Every 3 weeks, they will undergo a thorough assessment that includes:
  Symptom Assessment Nutritional Assessment (using NRS 2002 and PG-SGA) Psychological Assessment (using DT, GAD-7, FCR-7, ISI, PHQ-9)

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of enhanced follow-up with standard follow-up in postoperative patients with advanced gastric cancer who have undergone radical gastrectomy. The main questions it aims to answer are:

Can enhanced follow-up alleviate symptom burden and improve quality of life? What is the impact of enhanced follow-up on overall survival rates at 3 and 5 years post-surgery?

Participants will:

Be randomly assigned to either the enhanced follow-up group or the standard follow-up group.

Undergo comprehensive symptom, nutritional, and psychological assessments every 3 weeks (enhanced follow-up group).

Receive routine postoperative follow-up including medical examinations and treatments as needed, with additional assessments only when necessary (standard follow-up group).

Researchers will compare the enhanced follow-up group with the standard follow-up group to see if enhanced follow-up can improve quality of life and increase overall survival rates at 3 and 5 years post-surgery.

Outcomes will be measured using the EORTC QLQ-C30 quality of life questionnaire and overall survival rates. This prospective, single-center, randomized controlled clinical trial will span 5 years from the approval by the institutional ethics committee and will include 158 patients.

DETAILED DESCRIPTION:
1. Study Design and Methods 1.1 Study Design: This study is designed as a randomized controlled trial, with randomization implemented through an online clinical database. In this study, "enhanced follow-up" refers to comprehensive assessments every 3 weeks post-surgery, including symptom, nutritional, and psychological evaluations. "Standard follow-up" follows routine clinical practice, providing assessments only when necessary.

Experimental Group (Enhanced Follow-up Group) 1) Patients will undergo comprehensive assessments every 3 weeks post-surgery. 2) Nutritional Assessment: Using internationally recognized tools such as NRS 2002 and PG-SGA.

3) Psychological Assessment: Using tools such as the Distress Thermometer (DT), Generalized Anxiety Disorder 7-item scale (GAD-7), Fear of Cancer Recurrence 7-item scale (FCR-7), Insomnia Severity Index (ISI), and the Patient Health Questionnaire 9-item depression scale (PHQ-9).

Control Group (Standard Follow-up Group)

1. Patients will receive standard postoperative follow-up, including medical examinations and treatments as needed.
2. Nutritional and psychological assessments will be conducted only when deemed necessary by the patient or the healthcare provider.

For all patients, quality of life will be assessed using the EORTC QLQ-C30 questionnaire from 4 weeks post-surgery, every 6 weeks until 6 months post-chemotherapy. Additionally, 3-year and 5-year overall survival rates will be used to evaluate patient prognosis. Adverse events will be monitored and recorded, and treatment strategies will be adjusted as needed to ensure patient safety and study efficacy.

1.2 Nutritional Intervention

1.2.1 Nutritional Assessment Protocol:

Nutritional risk screening and comprehensive nutritional assessment will be conducted by dietitians, including Nutritional Risk Screening 2002 (NRS 2002), Patient-Generated Subjective Global Assessment (PG-SGA), dietary habits, and blood tests. Based on scores and clinical data, patients will be categorized into three groups:

1. Good nutrition or mild malnutrition group: Dietary guidance without delaying chemotherapy, with weekly nutritional risk screening.
2. Moderate malnutrition group: Dietary counseling and enteral nutrition support without delaying chemotherapy.
3. Severe malnutrition group: Counseling and nutrition support for 1-2 weeks before starting cancer treatment, continuing nutrition support during treatment.

NRS 2002: Includes disease score, nutritional impairment score, and age score, recommended by ESPEN and CSPEN for hospitalized patients. Patients are classified as at nutritional risk (score ≥ 3) or not at risk (score < 3).

PG-SGA: Designed for cancer patients, includes self-reported questionnaire and clinical assessment, with scores categorized as well-nourished (0-1), suspected malnutrition (2-3), moderate malnutrition (4-8), and severe malnutrition (≥9). In this study, NRS 2002 ≥ 3 or PG-SGA ≥ 4 indicates need for nutritional intervention.

1.2.2 Nutritional Support Protocol:

1. Development of Nutritional Support Plan: Based on the "Chinese Medical Association Guidelines for Parenteral and Enteral Nutrition" and individual clinical cases.
2. Nutritional Supply Standards: Target daily nutritional intake (including diet and parenteral/enteral nutrition support) set at 20-30 kcal/kg and 1-1.5 g/kg protein based on standard body weight.
3. Preference for Enteral Nutrition: Unless unable to achieve 60% target energy intake within 7 days, enteral nutrition is preferred; patients with contraindications should receive total parenteral nutrition.
4. Enteral Nutrition Formulation: Nutrison is the preferred formula. For intolerance or chronic disease complications, appropriate formulas such as Leskon or Abbott's Glucerna will be selected.
5. Calculation of Enteral Nutrition Support Level: If oral intake is reduced by 1/3-1/2, provide 2-3 cups/day (400-600 kcal) orally or via tube feeding. If reduced by more than 1/2, provide 3-5 cups/day (600-1000 kcal).
6. Preparation and Administration of Enteral Nutrition: Mix 9 scoops of Nutrison in 180 ml of warm water to make 1 cup of 1.0 kcal/ml nutritional solution, administered in divided doses (50-200 ml) daily. Initial volume should be half the prescribed amount, gradually increasing based on tolerance. Follow instructions for other brands.
7. Gradual Reduction or Discontinuation of Enteral/Parenteral Nutrition: When oral intake and enteral nutrition support meet 60% of nutritional needs, gradually reduce or discontinue support.

1.2.2 Indications for Discontinuing Nutritional Support:

1. Severe complications or contraindications to enteral nutrition.
2. Normal oral intake meeting daily nutritional needs.
3. Patient condition worsens, hemodynamic instability, or other contraindications.

1.2.4 Evaluation of Nutritional Support Effectiveness: Nutritional follow-up: The Nutritional Support Team (NST) will track patients' nutritional status every 3-4 weeks and adjust plans based on updates and tolerance until chemotherapy completion. Follow-up includes dietary and nutritional intake, weight changes, gastrointestinal symptoms or complications, and laboratory tests (serum electrolytes, liver/kidney function, blood glucose, lipids). Data will be recorded in case report forms (CRFs).

1.3 Psychological Intervention 1.3.1 Psychological Assessment Protocol:

1. Distress Thermometer (DT): A single-item scale from 0 (no distress) to 10 (extreme distress). The problem list covers five areas: practical, communication, emotional, physical, and spiritual/religious problems. A score ≥ 4 indicates high psychological distress.
2. Generalized Anxiety Disorder 7-item scale (GAD-7): Contains 7 items to assess the frequency of anxiety symptoms over the past two weeks, ranging from 0 (not at all) to 3 (nearly every day). A total score of 21, with scores ≥ 10 indicating possible clinically significant anxiety.
3. Fear of Cancer Recurrence 7-item scale (FCR-7): Specifically assesses the fear of cancer recurrence in survivors, with scores ranging from 0 (not at all) to 4 (a lot). A total score of 28, with higher scores indicating greater fear and potential need for professional support.
4. Insomnia Severity Index (ISI): Contains 7 items to evaluate insomnia severity, its impact on daily functioning, and the patient's perception of insomnia. Scores range from 0 (no problem) to 4 (very severe), with total scores ≥ 15 indicating severe insomnia.
5. Patient Health Questionnaire-9 (PHQ-9): Assesses depression severity over the past two weeks, with scores ranging from 0 (not at all) to 3 (nearly every day). A total score of 27, with higher scores indicating more severe depression.

1.3.2 Psychological Intervention Plan:

Assessments will be conducted every 3-4 weeks post-gastrectomy until 6 months post-surgery. Psychologists will help patients cope with the psychosocial impact of cancer treatment and provide further counseling as needed for patients and their family members.

1.3.2 Psychological Intervention:

1. Family Therapy: Interventions include "exploring family cohesion," "communicating thoughts and feelings," and "managing family conflicts." Typically involves three stages: 1) Identifying specific family issues and developing solutions; 2) Actual intervention; 3) Summary of psychological intervention. Frequency and duration of interventions will be adjusted based on each family's needs.
2. Individual Therapy: Principles include individualized psychological interventions based on clinical practice guidelines, with additional individual therapy provided during family interventions for those needing extra support.
3. Psychopharmacological Intervention: For patients meeting psychiatric diagnostic criteria (ICD-10 and DSM-IV), relevant psychopharmacological interventions (for anxiety, depression, insomnia, and adjustment disorders) will be provided. Medication will be offered to both intervention and control groups as deemed necessary by patients, family members, or attending physicians.

2. Withdrawal/Early Termination Criteria

Patients may voluntarily withdraw from the study at any time. Investigators may also decide to withdraw patients based on specific circumstances and medical judgment, ensuring the best interests of the patients. Reasons for withdrawal include:

1. Voluntary Withdrawal: Participants may withdraw at any time without providing a reason.
2. Non-compliance: Participants failing to adhere to study requirements, such as missing follow-ups or not completing necessary questionnaires.
3. Adverse Events: Occurrence of severe adverse events or other health issues related to the study, determined by the research doctor to be in the participant's best interest.
4. Disease Progression: Significant worsening of the participant's disease, preventing continued study participation.
5. Other Medical Reasons: Based on medical judgment, the research doctor determines that continuing participation is not suitable.
6. Loss to Follow-up: Participants lost to follow-up during the study, preventing further monitoring.

3. Exclusion Criteria

1. Patients not completing the scheduled treatment plan or follow-up.
2. Incomplete efficacy evaluation data, preventing effective assessment.
3. Efficacy evaluation not conducted as per the planned protocol, affecting result accuracy.
4. Non-compliance and termination cases should be followed up and analyzed according to the "intention-to-treat" (ITT) principle.

4. Follow-up Plan Establish a dedicated follow-up mechanism. Follow-up requirements: Every 3 months for the first 2 years post-surgery, then every 6 months until study completion. Follow-up includes lab tests (blood count, liver/kidney function, tumor markers), imaging (chest X-ray or CT, abdominal CT scan + enhancement, neck and supraclavicular lymph node ultrasound), and annual endoscopic examinations.

5. Follow-up Endpoints

1. Patient withdraws from the study.
2. Change in treatment due to complications or other conditions.
3. Patient death due to various causes.
4. Completion of the study period.
5. Loss to follow-up due to various reasons.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 72 years at the time of informed consent.
* Underwent radical total gastrectomy.
* Postoperative pathology confirmed advanced adenocarcinoma of the stomach or gastroesophageal junction.
* Estimated survival time ≥3 months.
* Good cognitive and reading abilities, capable of completing questionnaires.
* Willing and able to provide written informed consent for the study.

Exclusion Criteria:

* Participation in another clinical trial within 4 weeks prior to enrollment.
* Patients with other malignancies.
* Clinically significant cardiovascular disease, such as heart failure (NYHA III-IV), uncontrolled coronary artery disease, cardiomyopathy, arrhythmia, or hypertension.
* Neurological or psychiatric disorders affecting cognitive function, including central nervous system metastasis.
* Active infectious diseases, such as active hepatitis or tuberculosis.
* Uncontrolled systemic diseases, such as poorly controlled diabetes.
* Interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or evidence of interstitial lung disease on baseline chest X-ray/CT.
* Pregnant or breastfeeding.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Improvement | Assessed every 6 weeks from the 4th week post-surgery until 6 months post-chemotherapy completion.
  Measurement of quality of life improvement in postoperative advanced gastric cancer patients using the EORTC QLQ-C30 questionnaire. The assessment will include various dimensions such as physical functioning, emotional well-being, social functioning, and overall health status.

SECONDARY OUTCOMES:
3-Year Overall Survival Rate | 3 years post-surgery.
  The proportion of patients who are still alive 3 years after surgery.
5-Year Overall Survival Rate | 5 years post-surgery.
  The proportion of patients who are still alive 5 years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Xu, MD, PHD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in the article, after de-identification (text, tables, figures, and appendices), will be shared. This data will be made available to other researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 12 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal will be able to access the data. Proposals should be directed to the primary investigator. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Brown KW, Levy AR, Rosberger Z, Edgar L. Psychological distress and cancer survival: a follow-up 10 years after diagnosis. Psychosom Med. 2003 Jul-Aug;65(4):636-43. doi: 10.1097/01.psy.0000077503.96903.a6. PMID 12883115
- [Background] Guideline Committee of the Korean Gastric Cancer Association (KGCA), Development Working Group & Review Panel. Korean Practice Guideline for Gastric Cancer 2018: an Evidence-based, Multi-disciplinary Approach. J Gastric Cancer. 2019 Mar;19(1):1-48. doi: 10.5230/jgc.2019.19.e8. Epub 2019 Mar 19. No abstract available. PMID 30944757
- [Background] Lordick F, Carneiro F, Cascinu S, Fleitas T, Haustermans K, Piessen G, Vogel A, Smyth EC; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Gastric cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2022 Oct;33(10):1005-1020. doi: 10.1016/j.annonc.2022.07.004. Epub 2022 Jul 29. No abstract available. PMID 35914639
- [Background] Poulsen GM, Pedersen LL, Osterlind K, Baeksgaard L, Andersen JR. Randomized trial of the effects of individual nutritional counseling in cancer patients. Clin Nutr. 2014 Oct;33(5):749-53. doi: 10.1016/j.clnu.2013.10.019. Epub 2013 Nov 8. PMID 24269077
- [Background] Andrew IM, Waterfield K, Hildreth AJ, Kirkpatrick G, Hawkins C. Quantifying the impact of standardized assessment and symptom management tools on symptoms associated with cancer-induced anorexia cachexia syndrome. Palliat Med. 2009 Dec;23(8):680-8. doi: 10.1177/0269216309106980. Epub 2009 Oct 1. PMID 19797339
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Lu Z, Fang Y, Liu C, Zhang X, Xin X, He Y, Cao Y, Jiao X, Sun T, Pang Y, Wang Y, Zhou J, Qi C, Gong J, Wang X, Li J, Tang L, Shen L. Early Interdisciplinary Supportive Care in Patients With Previously Untreated Metastatic Esophagogastric Cancer: A Phase III Randomized Controlled Trial. J Clin Oncol. 2021 Mar 1;39(7):748-756. doi: 10.1200/JCO.20.01254. Epub 2021 Jan 8. PMID 33417481
- [Background] Baldwin C, Spiro A, Ahern R, Emery PW. Oral nutritional interventions in malnourished patients with cancer: a systematic review and meta-analysis. J Natl Cancer Inst. 2012 Mar 7;104(5):371-85. doi: 10.1093/jnci/djr556. Epub 2012 Feb 15. PMID 22345712